CLINICAL TRIAL: NCT04660136
Title: Usefulness of Contrast-enhanced Ultrasound (CEUS) in Crohn's Disease Pediatric Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2020-1010
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Crohn's Disease in Pediatric Patient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEUS (Experimental)
  Interventions: Biological: contrast enhanced ultrasound

INTERVENTIONS:
Biological: contrast enhanced ultrasound — We injected the second generation, ultrasonic contrast agent (SonoVue, Bracco, Milan, Italy) as a bolus of 0.03 ml/kg through a three-way 20-gauge catheter in an antecubital vein, followed by a bolus of 5 ml saline solution (0.9% NaCl).CEUS was performed with a 7.5MHz linear probe and contrast-tuned technology, based on allow mechanical index and a real-time scan to ensure the preservation of the contrast agent. A low acoustic power setting was used, expressing a low mechanical index (MI), 0.09-0.14, of a 7.5 MHz linear probe.

SUMMARY:
Purpose:

There is no previous contrast enhanced ultrasound (CEUS) study for pediatric Crohn disease patients. There are adult studies which included adolescent patients. More pediatric patients have been diagnosed as Crohn disease due to dietary change in Korea and it would be cost effective and clinically useful if CEUS was available in Crohn disease patients as a diagnostic and follow up tool.

Objective, hypothesis:

* Primary Objective To prospectively examine the feasibility of Contrast Enhanced Ultrasound (CEUS) in the assessment of Crohn's disease (CD) using endoscopy as a reference standard Feasibility was defined as the successful examination in over 90% of included patients.
* Secondary Objective To reaffirm the dosing and safety of ultrasound contrast agent and assess the image quality of the CEUS

Methodology:

This is a single center prospective observational study. Pediatric patients who was first diagnosed as CD with colonoscopy are enrolled in this study, The disease activity, clinical symptoms are also investigated. Within a period of maximally two weeks from the reference ileocolonoscopy and before any therapeutic changes, the patients underwent CEUS. CEUS was performed by one different pediatric radiologist, masked to all other imaging, endoscopic, and clinical data, except diagnosis of CD. CEUS was analyzed using quantification soft-ware (Vuebox), based on ROI at the most enhanced part of the bowel wall, quantitative parameters were calculated. After the first CEUS, CEUS would be performed after one year.

Pediatric population , 20 patients.

Imaging procedure:

Within a period of maximally two weeks from the reference ileocolonoscopy and before any therapeutic changes, the patients underwent CEUS on the same day. All studies started with a grey scale US examination to find the terminal ileum and assess wall thickness, induration of surrounding fatty tissue and enlarged lymphnodes. Stenosis and length of the pathologic bowel wall was estimated, as well as complications such as abscess formation and fistulae. The thickest segment of the terminal ileum was identified and used to perform analysis of contrast enhancement. The investigators injected the second generation, ultrasonic contrast agent (SonoVue, Bracco, Milan, Italy) as a bolus of 0.03 ml/kg through a three-way 20-gauge catheter in an antecubital vein, followed by a bolus of 5 ml saline solution (0.9% NaCl).CEUS was performed with a 7.5MHz linear probe and contrast-tuned technology, based on allow mechanical index and a real-time scan to ensure the preservation of the contrast agent. A low acoustic power setting was used, expressing a low mechanical index (MI), 0.09-0.14, of a 7.5 MHz linear probe. To assess the vascularization of the involved bowel loop, the contrast uptake over quantitative analysis of the brightness intensity was measured over a period of 40 s, in regions of interest (ROI) located manually in the intestinal wall with at least 2 cm2. The investigators used a dedicated software (Vuebox) and a time-intensity curve was automatically acquired. The quantitative measurement of the contrast uptake was obtained as the difference between the maximum enhancement value and the baseline value before the arrival of contrast.

Analysis, evaluation, reporting of results:

1. data acquisition: age, sex, initial treatment,

   - define involved bowel segment (5 segments: the terminal ileum, right colon (cecum and ascending), transverse colon, left colon (descending and sigmoid) and rectum), Gray scale US parameters identification of the terminal ileum, wall thickness measurement at the maximal diameter of the affected terminal ileum (pathological mural thickening defined as a wall thickness above 3 mm), evaluation of the affected bowel length, stratified wall appearance, perivisceral findings such as creeping fat and stenosis, fistula or abscess CEUS quantitative parameters, Numerous CEUS quantitative perfusion parameters can be derived from this curve. FT indicates fall time; mTTl, mean local transit time; PE, peak enhancement; RT, rise time; TTP, time to peak; WiAUC, wash-in area under the curve; WiR, wash-in rate; WiWoAUC, wash-in 1 wash-out area under the curve; WoAUC, wash-out area under the curve; and WoR, wash-out rate.

   Clinical and laboratory parameters (CDAI,, CRP, ESR and Calprotectin)
2. interpretation: independent interpretation of CEUS with colonoscopy as gold standard
3. outcome assessment

   * Successfully complete event number without adverse events
   * Treatment response: assessed by pediatric gastroenterologist by lab results, colonoscopy results, and patient symptom improvement

ELIGIBILITY:
Inclusion Criteria:

* Patients who are under the age of 18
* Patients who have Crohn's disease with colonoscopy from 2020.01-2022.02 in Severance Children Hospita

Exclusion Criteria:

* Patients who are over the age of 18 and under the age of two
* Patients who have other bowel disease or mass than Crohn's disease
* High allergic sensitivity to Sonovue injection agent or sulfur hexafluoride
* Patients who have right to left shunt, pulmonary hypertension, or systemic hypertension
* Patients who have end stage renal or liver disease or septic shock

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
feasibility of Contrast Enhanced Ultrasound (CEUS) in the assessment of Crohn's disease (CD) using endoscopy as a reference standard | 1 day
  Feasibility was defined as the successful examination in over 90 percent of included patients.

CONTACTS AND LOCATIONS:
Overall Officials: Haesung Yoon, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No